CLINICAL TRIAL: NCT04275999
Title: Epidermal Permeability Barrier Function and Stratum Corneum Hydration of Rosacea Following Application of Ivermectin
Brief Title: Rosacea and Ivermectin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00062694
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: The project will consist of a trial in which thirty subjects with rosacea receive ivermectin therapy and are randomized to receive either no intervention, a weekly digital survey to assess the subject's attitudes towards ivermectin therapy, or a portal hydration measurement device that measures TEWL rates and SC hydration levels. The study team will measure adherence objectively in all groups with electronic monitors attached to the containers of the ivermectin, which all subjects will be told to use daily for maintenance therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Control Group (Other): In the control group, all subjects will receive ivermectin equipped with an electronic monitor to measure adherence for daily treatment of rosacea. Subjects will not receive any follow-up intervention from the study team.
  Interventions: Drug: ivermectin
- Digital Interaction Group (Experimental): The digital interaction group will receive a survey by email each week asking about their use ivermectin generated by Causa Research; in addition to receiving ivermectin equipped with an electronic monitor to measure adherence for daily treatment of rosacea.
  Interventions: Drug: ivermectin; Behavioral: digital interaction
- GPSkin group (Experimental): The GPSkin group will receive the GPSkin Barrier® to measure their moisture level of their face daily. Subjects will be instructed to use the ivermectin once daily. Subjects also are receiving the ivermectin equipped with an electronic monitor to measure adherence for daily treatment of rosacea.
  Interventions: Drug: ivermectin; Device: GPSkin

INTERVENTIONS:
Drug: ivermectin — Subjects will be given the ivermectin with an electronic monitoring device attached with a return appointment at month 3 for end of study visit. Subjects will be instructed to use the ivermectin once daily.
Behavioral: digital interaction — Subjects will receive weekly digital interaction; an electronic survey asking about their use of the ivermectin which will have the electronic monitoring device attached. Subjects will be instructed to use the ivermectin once daily. They will have a 3 month return appointment for end of study visit.
  Other Names: digital interaction survey with ivermectin
  Arms: Digital Interaction Group
Device: GPSkin — Subjects in the GPSkin group will receive the GPSkin Barrier® to measure their moisture level of their face daily. Subjects will be instructed to use the ivermectin with the electronic monitoring device once daily. They will be scheduled for a 3 month end of study visit.
  Other Names: GPSkin Barrier®
  Arms: GPSkin group

SUMMARY:
The primary hypothesis is that weekly digital interactions and routine measurement of TEWL rates and SC hydration levels will promote patient adherence to maintenance ivermectin therapy and prevent disease relapse. The project will consist of a trial in which thirty subjects with rosacea receive ivermectin therapy and are randomized to receive either no intervention, a weekly digital survey to assess patient's attitudes towards ivermectin therapy, or a portal hydration measurement device that measures TEWL rates and SC hydration levels. The study team will measure adherence objectively in all groups with electronic monitors attached to the containers of the ivermectin, which all subjects will be told to use daily for maintenance therapy. Additionally, the hydration measurement device can transmit data to an Internet server via a smartphone using Bluetooth technology, thereby allowing providers to monitor a patient's TEWL rate and SC levels.

DETAILED DESCRIPTION:
Subjects will be offered an opportunity to participate in the study. Subjects will either have a diagnosis of rosacea. A total of 30 subjects will be enrolled. After consent and basic demographics, a study team member will use the GPSkin Barrier® to measure the baseline moisture level of the face of all subjects. Subjects will also fill out questionnaires pertaining to quality of life, accountability, and severity of rosacea.

Subjects will be randomized into one of three arms: the control group (n= 10), the digital interaction group (n=10), or the GPSkin group (n=10). All subjects will receive ivermectin equipped with an electronic monitor to measure adherence for daily treatment of rosacea. The digital interaction group will receive a survey by email each week asking about their use ivermectin generated by Causa Research. The subjects in the GPSkin group will receive the GPSkin Barrier® to measure their moisture level of their face daily. Subjects will be instructed to use the ivermectin once daily. Subjects will return at 3 Months. At this visit, the data from the electronic adherence monitoring will be downloaded, the ivermectin will be weighed, and the subject will fill out the same questionnaires (quality of life, accountability, and severity of rosacea). The intervention subjects will be evaluated on their use of the GPSkin Barrier® to measure their stratum corneum hydration. Subjects not randomized to the email intervention group will receive an accountability questionnaire at the beginning and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older.
* Subject has a working knowledge of English.
* Subject with a diagnosis of Rosacea
* Subjects without a known allergy to ivermectin
* Subjects with access to a smart phone

Exclusion Criteria:

* Subjects under 18 years of age.
* Subject does not have a working knowledge of English.
* Subject with a diagnosed skin condition other than rosacea
* Subjects with a known allergy to ivermectin
* Subjects without access to a smart phone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Adherence - MEMs Cap | Month 3
  Electronic monitoring of the ivermectin
Adherence - Drug Weight | Baseline
  the ivermectin will be weighed
Adherence - Drug Weight Change | Change from baseline to Month 3
  the ivermectin will be weighed
Transepidermal water loss (TEWL) rates | Baseline
  Use of the GPSkin Barrier device a portable hydration measurement device that measures TEWL rates
Transepidermal water loss (TEWL) rates | Change from baseline to 3 months
  Use of the GPSkin Barrier device a portable hydration measurement device that measures TEWL rates
Level of stratum corneum (SC) hydration | Baseline
  Use of the GPSkin Barrier device a portable hydration measurement device that measures TEWL rates
Level of stratum corneum (SC) hydration. | Change from baseline to 3 month
  Use of the GPSkin Barrier device a or a portable hydration measurement device that measures TEWL rates

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Health Sciences Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided